CLINICAL TRIAL: NCT04604977
Title: Feasibility and Effectiveness of Home-behavioral Program for Adolescents With Chronic Migraine and High Frequency Migraine Without Aura After the Covid-19 Emergency
Brief Title: Feasibility and Effectiveness of Home-behavioral Program for Adolescents With Migraine
Acronym: Be-Home-Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Be-Home-Kids
Record Dates: First submitted 2020-10-20; First posted 2020-10-27 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Headaches Chronic
MeSH Terms: conditions — Headache Disorders | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindfulness by Smartphone (Other): an approach that is alternative to current practice, particularly as far as reducing face-to-face hospital visits taking advantage of facilities offered by new technologies, besides including innovative and emerging treatment choices, namely a behavioural approach base on mindfulness
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Patients are followed with a standardized program including: education and support for behavioral measures, behavioral sessions, by mindfulness, once per week for 45 minutes for 6 weeks which usually delivered in groups of 4 - 8 patients.

SUMMARY:
Chronic Migraine and Migraine without aura at high frequency are disabling conditions also in adolescence age (2% of adolescents report chronic migraine) Common pharmacological treatments are often inadequate. It has been reported that clinical results can be improved when traditional therapies are combined with behavioral approaches in particular mindfulness, that help patients to become more conscious about their symptoms and able to manage pain without medication. Generally, according to standard clinical practice, young patients (12-17 yrs old) treated by mindfulness practice come to the hospital to practice mindfulness in small groups of patients for 6 weekly 45 minutes sessions. As the emergency situation due to the Corona-virus pandemic phenomenon in Italy, patients missed the possibility to come for the regular practice to the hospital: for this reason the investigators propose a small pilot study to enforce the use of technology for patients so that they can continue to be followed during their therapeutic process. This preliminary study will be conducted on 25 patients They will be trained to practice mindfulness daily by a standard session of 12 minutes on their smartphone recorded by the expert who generally manage their sessions at the hospital. Also a weekly video-session will be performed to evaluate the clinical condition, to practice guided mindfulness sessions and to encourage to use strategies for pain management . This modality will allow patients to continue their therapeutic process and to be followed regularly during the one year after treatment. Follow up sessions are planned every three months: these meetings at the hospital will be face-to-face with every patient to check the clinical condition by the patient's diary. Last follow up one year after treatment.

DETAILED DESCRIPTION:
Background and significance Chronic Migraine is not so unusual in pediatric and adolescent age and is about 2% of population in adolescent age. The literature of the last decades confirmed the need to taking care of these patients susceptible to develop medication overuse. There are different pharmacological treatments for migraine in young patients but no one of them has specific indication for this category of patients and their efficacy reaches 30/40% leaving many side effects difficult to manage at this age. The feasibility and the effectiveness of behavioral approaches has been already documented in clinical experiences of the last decades: these approaches revealed efficacy in long-term studies and with control groups and they are totally free of unpleasant effects. Mindfulness practice is one of the most recent behavioral approaches that combined with Acceptance Commitment Therapy offer a suitable and adequate treatment for adolescent patients. These approaches make patients more conscious about their problem and able to learn techniques alternative to medications for managing pain.. Mindfulness and other behavioral therapies have done significant results in terms of clinical improvement for these patients and they are well accepted with a high adherence level. This preliminary study will be performed considering that the Covid-19 emergency reduced significantly the possibility for patients to follow sessions at the hospital and to move among the different Italian regions and the investigators organized a program with education and support by mindfulness , delivered by video sessions. According to the protocols at the Headache Center of the Besta Institute in Milan Italy, patients of this category are followed with a standardized program including: education and support for behavioral measures, behavioral sessions, by mindfulness, once per week for 45 minutes for 6 weeks which usually delivered in groups of 4 - 8 patients. This approach may be particularly useful in helping patients to obtain a better outcome. All the above discussed considerations are even more relevant in this emergency situation due to the Corona-virus pandemic phenomenon in Italy, with its consequences on mobility of patients and clinical practice. In order to promote different modalities to respond to the needs of patients suffering from this disabling condition during the emergency, exercise-based telemedicine and smartphone applications seem very appropriate, as they have been recently tested in the management of chronic pain conditions. This preliminary study will be performed considering that the Covid-19 emergency reduced significantly the mobility of patients, particularly those living in other Italian regions than Lombardy, and in view of providing an effective and somewhat innovative treatment program for this class of patients. The proposed treatment intervention is based on investigators' experience, and on published reports, but it specifically includes a home based program, visits performed as Video calls, and educational and support strategies aimed to develop skills to reduce clinical symptoms and to cope with pain by a standardized behavioural approach based on mindfulness -

which will be delivered mainly by telemedicine and smartphone applications . The aim of this pilot study is to assess the feasibility and the effectiveness at long-term on relevant outcomes of a specific protocol, designed to be appropriate during the emergency situation due to COVID-19 epidemic, by an approach that is alternative to current practice, particularly as far as reducing face-to-face hospital visits taking advantage of facilities offered by new technologies, besides including innovative and emerging treatment choices, namely a behavioural approach base on mindfulness

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Chronic Migraine or High Frequency Migraine without aura
* written informed consent

Exclusion Criteria:

* co-existent severe medical or psychiatric illnesses, documented by specific previous diagnoses
* seizures
* use of opioids
* participation to other projects with behavioral approaches in the last

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
reduction of headache days | at 6 months and 12 months follow-up compared with baseline (Headache Daily Diary)
  reduction of at least 50 % of headache days during the treatment period

SECONDARY OUTCOMES:
reduction of headache days until last follow up | at 12 months from withdrawal program (assessed by Daily Diary Card)
  reduction of at least 50 % of headache days until the last follow up (assessed by Daily Diary Card)
disability score | 6 months - 12 months
  decrease in disability score (Ped MIDAS) - (score of PedMIDAS: 0-10 little disability; 11-30 mild disability; 31-50 moderate disability; more than 50 severe disability)
catastrophising attitude | 6 months - 12 months
  decrease in catastrophising attitude (PCS) - Score more than 30 : clinically relevant level of catastrophising
depression symptoms | 6 months - 12 months
  decrease in depression symptoms (Kovacs) - score =15 mild depression; 15-20 moderate depression; more than 25 severe depression);
trait-state anxiety symptoms (STAI X1-X2) | 6 months - 12 months
  decrease in trait-state anxiety symptoms (STAI X1-X2) - score more than 40 anxiety symptoms abnormal

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Neuroalgology Unit, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided